CLINICAL TRIAL: NCT00078520
Title: Treatment of Chronic Lymphocytic B-Leukemia (B-CLL) With Human IL-2 and CD40 Ligand and Plasmid Gene Modified Autologous Tumor Cells (CLIPA)
Brief Title: Treatment of B-CLL With Human IL-2 and CD40 Ligand and Plasmid Gene Modified Autologous Tumor Cells
Acronym: CLIPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Dist Serv Prof, Center for Gene Therapy, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11967; CLIPA
Record Dates: First submitted 2004-03-01; First posted 2004-03-02 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Leukemia; Leukemia, B-Cell, Chronic
Keywords: Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 (Experimental): Patients may be treated with a minimum of 3-6 injections of their IL-2-secreting and CD40L-expressing autologous B-CLL cells, separated by one to two weeks in an immunological treatment window. Any patient whose disease regresses after the administration of 6 injections may be offered further injections (i.e. more than 6 injections) of tumor vaccine at the dose level previously administered, if enough vaccines are available. Patients will receive a fixed dose of IL-2 secreting B-CLL cells throughout the entire treatment protocol while an escalating number of CD40L-expressing B-CLL cells will be given at each dose-level.
  Interventions: Biological: Dose Level 1
- Dose Level 2 (Experimental): Patients may be treated with a minimum of 3-6 injections of their IL-2-secreting and CD40L-expressing autologous B-CLL cells, separated by one to two weeks in an immunological treatment window. Any patient whose disease regresses after the administration of 6 injections may be offered further injections (i.e. more than 6 injections) of tumor vaccine at the dose level previously administered, if enough vaccines are available. Patients will receive a fixed dose of IL-2 secreting B-CLL cells throughout the entire treatment protocol while an escalating number of CD40L-expressing B-CLL cells will be given at each dose-level.
  Interventions: Biological: Dose Level 2
- Dose Level- Fixed Dose (Experimental): Patients may be treated with a minimum of 3-6 injections of their IL-2-secreting and CD40L-expressing autologous B-CLL cells, separated by one to two weeks in an immunological treatment window. Any patient whose disease regresses after the administration of 6 injections may be offered further injections (i.e. more than 6 injections) of tumor vaccine at the dose level previously administered, if enough vaccines are available. Patients will receive a fixed dose of IL-2 secreting B-CLL cells throughout the entire treatment protocol while an escalating number of CD40L-expressing B-CLL cells will be given at each dose-level.
  Interventions: Biological: Dose Level 2- Fixed Dose

INTERVENTIONS:
Biological: Dose Level 1 — IL-2-B-CLL 2 x 10^7; CD40L-B-CLL 0
  Arms: Dose Level 1
Biological: Dose Level 2 — IL-2-B-CLL 2 x 10^7; CD40L-B-CLL 2 x 10^6
  Arms: Dose Level 2
Biological: Dose Level 2- Fixed Dose — IL-2-B-CLL 2 x 10^7; CD40L-B-CLL 2 x 10^7
  Arms: Dose Level- Fixed Dose

SUMMARY:
This study is for patients that have chronic lymphocytic leukemia (CLL). This research study aims to determine the safety and dosage of special cells that may make the patients own immune system fight the cancer.

To do this, we will put a special gene into cancer cells that have been taken from the patients body. This will be done in the laboratory. This gene will make the cells produce interleukin 2 (IL-2), which is a natural substance that may help the immune system kill cancer cells. Additionally, we will stimulate the cancer cells with another natural protein called CD40 ligand (CD40L), which experiments in animal and human cells in vitro demonstrated can help IL-2 perform better.

Some of these cells will then be put back into the patient's body. Studies of cancers in animals and in cancer cells that are grown in laboratories suggest that combining substances like IL-2 and CD40L helps the body kill cancer cells. An experimental treatment similar to this has already been used in children and similar experimental treatments are being used in adults with other cancers.

DETAILED DESCRIPTION:
This is a phase I trial to assess the safety of a dose escalation of hCD40L-expressing autologous tumor cells with a fixed dose of recombinant hIL-2 gene transduced autologous leukemic blasts. All eligible patients will be treated with a minimum of three and up to six injections. There will be no use of placebo or control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for administration of their vaccine if they present with B-CLL (not in Richters transformation) with (group A) or without (group B) (Inclusion of B-CLL) measurable disease. Untreated or complete remission patients will be enrolled for vaccine administration in a therapeutic (i.e., no chemotherapy) window of three months. If during these three months (necessary to complete the vaccine study), the patient presents with rapid clinical progression, he or she will be excluded from our current study and will receive treatment according to the standard institutional guidelines. IMPORTANT NOTE: vaccine production for complete remission patients can only be achieved if tumor cells have been collected BEFORE entering complete remission.
* Patients must have a life expectancy of at least 10 weeks.
* Patients must have ECOG performance status of 0-2 as below: 0 = up and about, no restriction, 1 = Ambulatory, no strenuous activity, 2 = Ambulatory, capable of self-care appropriate for age. Up and about > 50% of time, but unable to carry out any physical activities or attend school, 3 = Limited self-care only. Up and about < 50% of time, 4 = Disabled, no self care. Bedridden or confined to chair.
* Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study, and must have an absolute neutrophil count (ANC) of > / = 500/mL, absolute lymphocyte count (ALC) > / = 200/mL, hemoglobin > / = 8g/dL, and platelet count > / = 50,000/mL
* Patients must not be infected at time of protocol entry, and should not be receiving antibiotics (other than prophylactic trimethoprim sulfamethoxazole).
* Patients must be HIV-negative.
* Patients must be willing to practice appropriate birth control methods during the study and for 3 months after the study is concluded. This includes total abstinence, oral contraceptives, an intrauterine device, contraceptive implants under the skin, contraceptive injections (Depo-Provera). Contraceptive foam with a condom is allowed. The male partner should use a condom.
* Patients must not be suffering from an autoimmune disease (including active graft-versus-host disease-GvHD, refractory immune thrombocytopenia-ITP or refractory autoimmune hemolytic anemia-AIHA) and should not be receiving immunosuppressive drugs.
* Patients must have adequate liver function (total bilirubin < / = 1.5mg/dl, SGOT < / = 2 times normal, normal prothrombin time).
* Patients must have adequate renal function (creatinine less than 3 times normal for age or creatinine clearance > 80mg/min/1.73m2).
* Patients must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side-effects. Patients will be given a copy of the consent form.
* Patient must not have received treatment with other investigational agents within the last 4 weeks.

Exclusion Criteria:

* Richters transformation (aggressive non-Hodgkins lymphoma),
* active infection,
* significant autoimmune disease (including active GvHD, ITP and AIHA),
* requirement for immunosuppressive drugs,
* inadequate liver and/or renal function,
* pregnancy or lactation,
* refusal to practice birth control methods,
* seropositive for HIV,
* life expectancy less than 10 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
safety of injections of autologous malignant B cells from B-CLL patients, which have been modified to secrete hIL-2 and hCD40L. | 12 weeks

SECONDARY OUTCOMES:
anti-tumor immune responses | 15 years
obtain preliminary data on the anti-tumor effects of this treatment regimen. | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: MALCOLM K BRENNER, MD, Study Chair — Baylor College of Medicine
Locations (1):
- The Methodist Hospital, Houston, Texas, United States